CLINICAL TRIAL: NCT01173744
Title: Comparison of Gamma Nail Versus Dynamic Hip Screw for the Treatment of Unstable Intertrochanteric Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Dror Lakstein, MD, Wolfson MC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0076-10-WOMC
Record Dates: First submitted 2010-07-27; First posted 2010-08-02 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2010-07

CONDITIONS: Intertrochanteric Femoral Fractures
Keywords: Intertrochanteric femoral fractures - unstable

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Gamma-3 Nail (Experimental)
  Interventions: Device: Gamma-3 Nail
- DHS (Active Comparator)
  Interventions: Device: DHS

INTERVENTIONS:
Device: Gamma-3 Nail — Gamma-3 Nail (stryker)
  Arms: Gamma-3 Nail
Device: DHS — DHS (Zimmer)
  Arms: DHS

SUMMARY:
The objective of the study is to examine the treatment of unstable Intertrochanteric fractures with the short Gamma nail, compared to the use of the dynamic hip screw (DHS).

This is a prospective study. Sixty patients with unstable Intertrochanteric fractures will be randomized to be treated using either Gamma nail or DHS. The patients will be followed for 12 months. The primary endpoint is the clinical outcome as measured by the Merle d'Aubigne and Postelhip score.

ELIGIBILITY:
Inclusion Criteria:

* Acute Intertrochanteric fracture - A1-32 AO/OTA
* Abbreviated mental score >6
* Community ambulator (pre-fracture state)

Exclusion Criteria:

* Previous arthritis
* Pathological fracture
* Chronic corticosteroid use
* Concomitant lower extremity fractures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome as measured by the Merle d'Aubigne and Postel hip score | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- E. WOlfson medical center, Holon, Israel